CLINICAL TRIAL: NCT04558463
Title: The Effectivity and Safety of Favipiravir Compared to Oseltamivir as Adjuvant Therapy for COVID-19: An Open Label Trial
Brief Title: The Effectivity and Safety of Favipiravir Compared to Oseltamivir as Adjuvant Therapy for COVID-19
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Dante Saksono Harbuwono, Sp.PD, PhD, Principal Investigator, Head of Endocrinology Division, Department of Internal Medicine, Dr. Cipto Mangunkusumo National Referral Hospital, Faculty of Medicine Universitas Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-04-0455
Record Dates: First submitted 2020-09-03; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: COVID-19; Favipiravir; oseltamivir; adjuvant; effectivity
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; Oseltamivir

STUDY DESIGN:
Intervention Model Description: Subjects will be divided into two groups: favipiravir and oseltamivir as adjuvant therapy in addition to standard therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Experimental): The favipiravir group received loading dose and maintenance dose of Favipiravir for 2 up to 7 days in addition to standard therapy
  Interventions: Drug: Favipiravir
- Oseltamivir (Active Comparator): The oseltamivir group was given oseltamivir for 7 days.
  Interventions: Drug: Oseltamivir 75mg

INTERVENTIONS:
Drug: Favipiravir — The favipiravir group received loading dose of 1600 mg twice a day (3200 mg/day) on the first day and continued with 600 mg twice a day (1200 mg/day) for the next 2nd - 7th day in addition to the standard therapy.
  Standard therapy: administration of azithromycin 500 mg/day or levofloxacin 750 mg/day for 5 days, chloroquine (either Sulphur-based chloroquine 600 mg/day or chloroquine phosphate 100 mg/day or hydroxychloroquine 400 mg/day) for 5-7 days, vitamin C, oxygen therapy according to the patients clinical condition, comorbid therapy and other symptomatic treatment such as antipyretic drug
  Other Names: Avigan® (favipiravir)
  Arms: Favipiravir
Drug: Oseltamivir 75mg — The oseltamivir group was given twice a day of 75 mg of oseltamivir (150 mg/day) for 7 days in addition to standard therapy
  Standard therapy: administration of azithromycin 500 mg/day or levofloxacin 750 mg/day for 5 days, chloroquine (either Sulphur-based chloroquine 600 mg/day or chloroquine phosphate 100 mg/day or hydroxychloroquine 400 mg/day) for 5-7 days, vitamin C, oxygen therapy according to the patients clinical condition, comorbid therapy and other symptomatic treatment such as antipyretic drug
  Other Names: Oseltamivir
  Arms: Oseltamivir

SUMMARY:
This study aims to analyze the effectiveness and safety of Avigan® (favipiravir) compared to Oseltamivir as an adjuvant therapy among adult COVID-19 patients. This study will be conducted in a hospital setting, recruiting adult COVID-19 patients with mild, moderate, and severe symptoms. Subjects will be randomly given Favipiravir or Oseltamivir as an adjuvant therapy to standard COVID-19 treatment. Patients will be followed up for 21 days after the first dose of intervention given. The primary outcomes of this study are the improvement of radiology results and RT PCR negative conversion during follow up. The secondary outcomes are adverse events, hospital length of stay (LOS), and Case fatality rate (CFR)

DETAILED DESCRIPTION:
This open-label trial aims to analyze the effectiveness and safety of Avigan® (favipiravir) compared to Oseltamivir as an adjuvant therapy among adult COVID-19 patients. This study will be conducted in a hospital setting, recruiting adult COVID-19 patients with mild, moderate, and severe symptoms. Subjects will be randomly given Favipiravir or Oseltamivir as an adjuvant therapy to standard COVID-19 treatment. Patients will be followed up for 21 days after the first dose of intervention given. The primary outcomes of this study are clinical improvements determined by laboratory measurements and radiology results. The secondary outcomes are adverse events, hospital length of stay (LOS), and Case fatality rate (CFR)

ELIGIBILITY:
Inclusion Criteria:

1. adult patients aged 18-75 years old
2. Patients with COVID-19 showing symptoms and confirmed with positive RT PCR test AND OR COVID-19 IgM/IgG rapid test
3. No history of favipiravir or oseltamivir allergy
4. Consented to participate in the trial.

Exclusion Criteria:

1. Pregnant women
2. Breastfeeding mother
3. Patients with markedly elevated liver enzyme (ALT and/or AST) of more than three times from baseline level
4. Reduced kidney function with estimated glomerular filtration rate (eGFR) <30 mL/min OR serum creatinine > 2 mg/dL
5. Patients with history of heart failure
6. Tuberculosis infection that was treated with pyrazinamide
7. Asthma that was treated with theophylline
8. Type 2 diabetes that was treated with repaglinid

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Clinical radiologic changes | 14 days
  Changes of lung infiltrate in chest xray AND/OR GGO in chest CT scan after 14 days of follow up period This outcome measured will displayed as improvement/no changes/deterioration of radiologic examination results
Percentage of RT-PCR test convertion | 14 days
  Convertion of RT-PCR swab result from positive to negative at the end of 14 days study follow up This outcome measured will displayed as convertion OR no conversion

SECONDARY OUTCOMES:
Adverse event | 14 days
  Mild to moderate adverse event serious adverse event such as sever allergy and increased transaminase enzyme >3x normal limit
Hospital length of stay (LOS) | 14 days
  Days of hospitalization from the first dose of intervention
Case Fatality Rate (CFR) | 14 days
  CFR is calculated from mortality rate during hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Dante S Harbuwono, MD, PhD, Principal Investigator — Head of Division Endocrinology, Department of Internal Medicine, FMUI
Locations (1):
- Cipto Mangunkusumo National Referral Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No